CLINICAL TRIAL: NCT04570670
Title: A Single-Dose, Randomized, Open-Label, 2-Way Crossover, Comparative Bioavailability Study of BLS-11 (Monomethyl Fumarate) 190 mg and Tecfidera (Dimethyl Fumarate) 240 mg in Healthy Male and Female Subjects Under Fasting Conditions
Brief Title: Comparative Bioavailability of BAFIERTAM™ (Monomethyl Fumarate) and Tecfidera® (Dimethyl Fumarate) in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Banner Life Sciences LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BLS-11-104
Record Dates: First submitted 2020-09-22; First posted 2020-09-30 (Actual); Results first posted 2021-07-28 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-03

CONDITIONS: Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — monomethyl fumarate; Dimethyl Fumarate

STUDY DESIGN:
Intervention Model Description: Subjects were randomized to 1 of 2 treatment sequences prior to the first dose.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Test (BLS-11) (Experimental): A single oral dose administration of BLS-11 190 mg (2 × 95 mg monomethyl fumarate delayed-release capsules) at Hour 0 on Day 1
  Interventions: Drug: monomethyl fumarate 190 mg
- Reference (Tecfidera) (Active Comparator): A single oral dose administration of Tecfidera 240 mg (1 × 240 mg dimethyl fumarate delayed-release capsule) at Hour 0 on Day 1
  Interventions: Drug: dimethyl fumarate 240 mg

INTERVENTIONS:
Drug: monomethyl fumarate 190 mg
  Other Names: BAFIERTAM; BLS-11
  Arms: Test (BLS-11)
Drug: dimethyl fumarate 240 mg
  Other Names: Tecfidera
  Arms: Reference (Tecfidera)

SUMMARY:
The primary objective of this study was to assess the bioequivalence of the test product (Bafiertam; BLS-11; monomethyl fumarate) 190 mg versus Tecfidera® (dimethyl fumarate) 240 mg based on the Cmax and Area Under the Curve (AUC) values of monomethyl fumarate (MMF) determined after a single dose under fasting conditions.

DETAILED DESCRIPTION:
This was a single-dose, open-label, randomized, 2-way crossover study, evaluating the comparative pharmacokinetics of the test product (MMF) versus the reference product (DMF) under fasting conditions. Fifty (50) healthy, adult male and non-pregnant female subjects were enrolled. Screening of subjects occurred within 21 days prior to the first dose. Subjects were randomized to 1 of 2 treatment sequences prior to the first dose.

In each period, subjects received a single oral dose of MMF 190 mg administered as two 95 mg delayed-release capsules (test product) or Tecfidera® 240 mg DMF delayed-release capsule (reference product), followed by blood sampling (including predose samples) up to 24 hours postdose for the determination of plasma concentrations of MMF. There was a washout period of 2 days between the 2 doses.

Safety was monitored throughout the study by repeated clinical and laboratory evaluations.

ELIGIBILITY:
Inclusion Criteria:

1. Continuous non-smoker who had not used nicotine-containing products for at least 3 months prior to the first dose and throughout the study.
2. Body mass index (BMI) ≥ 18.5 and ≤ 29.9 kg/m2 at Screening.
3. Medically healthy as determined by the Investigator or designee with no clinically significant medical history, physical examination, laboratory profiles, vital signs or electrocardiograms (ECGs), as deemed by the Investigator or designee.
4. Females of childbearing potential: not pregnant and either sexually inactive (abstinent) for 14 days prior to the first dose and throughout the study or using one of the following acceptable birth control methods: hormonal oral contraceptives, vaginal ring, transdermal patch, or nonhormone or hormone releasing intrauterine device for at least 3 months prior to the first dose with either a physical (e.g., condom, diaphragm, or other) or a chemical (e.g., spermicide) barrier method from the time of Screening and throughout the study; depot/implantable hormone (e.g., Depo Provera®, Implanon®) for at least 3 months prior to the first dose and throughout the study.

   In addition, female subjects of childbearing potential were advised to remain sexually inactive or to keep the same birth control method for at least 7 days following the last dose.
5. Females of non-childbearing potential: had undergone one of the following sterilization procedures at least 6 months prior to the first dose: hysteroscopic sterilization; bilateral tubal ligation or bilateral salpingectomy; hysterectomy; bilateral oophorectomy or were postmenopausal with amenorrhea for at least 1 year prior to the first dose and follicle-stimulating hormone (FSH) serum levels consistent with postmenopausal status as per Investigator's or designee's judgment.
6. Non-vasectomized male subjects agreed to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days beyond the last dose of study drug. (No restrictions were required for a vasectomized male provided his vasectomy had been performed 4 months or more prior to the first dose of study drug. A male who had been vasectomized less than 4 months prior to the first dose of study drug, followed the same restrictions as a non-vasectomized male.)
7. Males agreed not to donate sperm from the first dose until 90 days after dosing.
8. Understood the study procedures in the Informed Consent Form (ICF), and were willing and able to comply with the protocol.

Exclusion Criteria:

1. Subject was mentally or legally incapacitated or had significant emotional problems at the time of the Screening visit or expected during the conduct of the study.
2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the Investigator or designee.
3. History of any illness that, in the opinion of the Investigator or designee, might have confounded the results of the study or posed an additional risk to the subject by their participation in the study.
4. History or presence of alcoholism or drug abuse within the past 2 years prior to the first dose.
5. History or presence of hypersensitivity or idiosyncratic reaction to the study drugs or related compounds.
6. Female subjects with a positive serum pregnancy test at Screening or Check-in, or who were lactating.
7. Positive urine drug, alcohol, or cotinine results at Screening or Check-in.
8. Positive results at Screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV).
9. Seated blood pressure was less than 90/40 mmHg or greater than 140/90 mmHg at Screening.
10. Seated heart rate was lower than 40 beats per minute (bpm) or higher than 99 bpm at Screening.
11. Abnormal 12-lead ECG deemed clinically significant by the Investigator or designee at Screening or prior to the first dose.
12. Unable to refrain from or anticipated the use of any drug, including prescription and non-prescription medications, or herbal remedies, beginning 14 days prior to the first dose and throughout the study. Medication listed as part of acceptable birth control methods was allowed. Hormone replacement therapy was also allowed. Acetaminophen (up to 2 g per 24-hour period) may have been permitted, as necessary during the study.
13. Had been on a diet incompatible with the on study diet, in the opinion of the Investigator or designee, within the 28 days prior to the first dose and throughout the study.
14. Donation of blood or significant blood loss within 30 days prior to the first dose.
15. Plasma donation within 7 days prior to the first dose.
16. Participation in another clinical study within 28 days prior to the first dose. The 28-day window was derived from the date of the last blood collection or dosing, whichever was later, in the previous study to Day 1 of Period 1 of the current study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2017-01-06 (Actual); Primary Completion 2017-02-17 (Actual); Study Completion 2017-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franck Rousseau, MD, Study Director — Banner Life Sciences LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lategan TW, Wang L, Sprague TN, Rousseau FS. Pharmacokinetics and Bioavailability of Monomethyl Fumarate Following a Single Oral Dose of Bafiertam (Monomethyl Fumarate) or Tecfidera(R) (Dimethyl Fumarate). CNS Drugs. 2021 May;35(5):567-574. doi: 10.1007/s40263-021-00799-9. Epub 2021 Mar 30. PMID 33797063
- See also: Open Access — https://rdcu.be/chVM1

RESULTS

PARTICIPANT FLOW:
Groups:
- Randomization Sequence AB: Treatment A: A single oral dose of BLS-11 190 mg (2 x 95 mg)
  Treatment B: A single oral dose of Tecfidera® 240 mg (1 × 240 mg)
- Randomization Sequence BA: Treatment B: A single oral dose of Tecfidera® 240 mg (1 × 240 mg)
  Treatment A: A single oral dose of BLS-11 190 mg (2 x 95 mg)
Period: Overall Study
Arm/Group | Randomization Sequence AB | Randomization Sequence BA
Started | 25 | 25
Completed | 24 | 25
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Randomization Sequence AB: Treatment A: A single oral dose of BLS-11 190 mg (2 x 95 mg) MMF
  Treatment B: A single oral dose of Tecfidera® 240 mg (1 × 240 mg) DMF
- Randomization Sequence BA: Treatment B: A single oral dose of Tecfidera® 240 mg (1 × 240 mg) DMF
  Treatment A: A single oral dose of BLS-11 190 mg (2 x 95 mg) MMF
- Total: Total of all reporting groups
Arm/Group | Randomization Sequence AB | Randomization Sequence BA | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.4 (9.85) | 38.0 (8.22) | 36.2 (9.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 19 | 17 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 12 | 27
  Not Hispanic or Latino | 10 | 13 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 19 | 19 | 38
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50
Weight [Mean (Standard Deviation); unit: kg] | 72.98 (9.450) | 74.78 (12.512) | 74.78 (11.011)
Height [Mean (Standard Deviation); unit: cm] | 168.6 (7.55) | 170.3 (10.58) | 169.5 (9.14)
Body Mass Index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 25.625 (2.4142) | 25.678 (2.9237) | 25.651 (2.6537)

OUTCOME MEASURES:

1. Primary Outcome: The Bioequivalent (BE) Comparison of AUC0-inf of Monomethyl Fumarate (MMF) Between Treatments
Description: Pharmacokinetics: Plasma concentrations of MMF will be determined and used to calculate AUC0-inf MMF for each treatment. Venous blood samples were collected immediately prior to dosing (time 0), and then 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 9, 10, 11, 12, and 24 hours postdose.
Time Frame: 24 hours
Population: One subject in the Reference (Tecfidera) group was excluded from AUC0-inf calculations because of missing or unreportable values and was excluded from the statistical analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- Test (BLS-11): A single oral dose administration of BLS-11 190 mg (2 × 95 mg monomethyl fumarate delayed-release capsules) at Hour 0 on Day 1
  monomethyl fumarate 190 mg
- Reference (Tecfidera): A single oral dose administration of Tecfidera 240 mg (1 × 240 mg dimethyl fumarate delayed-release capsule) at Hour 0 on Day 1
  dimethyl fumarate 240 mg
Arm/Group | Test (BLS-11) | Reference (Tecfidera)
Number analyzed (Participants) | 49 | 48
ng*hr/mL | 2984 (25.9) | 3116 (23.9)

2. Primary Outcome: The BE Comparison of Cmax of Monomethyl Fumarate (MMF) Between Treatments
Description: Pharmacokinetics: Plasma concentrations of MMF will be determined and used to calculate the Cmax of MMF for each treatment.Venous blood samples were collected immediately prior to dosing, and then 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 7.5, 8, 9, 10, 11, 12, and 24 hours postdose.
Time Frame: 24 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Test (BLS-11) | Reference (Tecfidera)
Number analyzed (Participants) | 49 | 49
ng/mL | 1760 (34.8) | 1680 (33.8)

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Test (BLS-11) | Reference (Tecfidera)
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/49
Other Adverse Events (participants affected / at risk) | 31/50 | 29/49
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test (BLS-11) (N=50) | Reference (Tecfidera) (N=49)
Palpitations (Cardiac disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 1
Chills (General disorders) | 1 | 0
Feeling Hot (General disorders) | 1 | 0
Vessel puncture site erythema (General disorders) | 0 | 1
Vessel puncture site pain (General disorders) | 0 | 1
Vessel puncture site swelling (General disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Euphoric mood (Psychiatric disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 1
Flushing (Vascular disorders) | 30 | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-12): https://cdn.clinicaltrials.gov/large-docs/70/NCT04570670/Prot_SAP_000.pdf